CLINICAL TRIAL: NCT07258849
Title: A Phase 1, Multicenter, Randomized, Placebo-Controlled, Investigator- and Participant-Blinded, Single- and Multiple-Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of LY4213663 in Healthy Participants, and Two Open-Label, Multiple-Dose Evaluations of LY4213663 in Patients With Rheumatoid Arthritis.
Brief Title: A Study of LY4213663 in Healthy Participants and Participants With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27749; 2025-523980-39-00 (EU CTIS Number); J6T-MC-KYAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LY4213663 (Part A) (Experimental): Single-ascending dose (SAD) of LY4213663 administered subcutaneously (SC) and intravenously (IV) in healthy participants
  Interventions: Drug: LY4213663
- Placebo (Part A) (Placebo Comparator): SAD placebo administered SC and IV
  Interventions: Drug: Placebo
- LY4213663 (Part B) (Experimental): Multiple-ascending doses (MAD) of LY4213663 administered SC and IV in healthy participants
  Interventions: Drug: LY4213663
- Placebo (Part B) (Placebo Comparator): MAD placebo administered SC and IV
  Interventions: Drug: Placebo
- LY4213663 (Parts C and D) (Experimental): Multiple doses of LY4213663 administered SC and IV in participants with RA
  Interventions: Drug: LY4213663

INTERVENTIONS:
Drug: LY4213663 — Administered SC
  Arms: LY4213663 (Part A); LY4213663 (Part B); LY4213663 (Parts C and D)
Drug: LY4213663 — Administered IV
  Arms: LY4213663 (Part A); LY4213663 (Part B); LY4213663 (Parts C and D)
Drug: Placebo — Administered SC
  Arms: Placebo (Part A); Placebo (Part B)
Drug: Placebo — Administered IV
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The purpose of this study is to evaluate how well LY4213663 is tolerated and what side effects may occur in healthy participants and participants with rheumatoid arthritis (RA). The study drug will be administered either subcutaneously (SC) (under the skin) or intravenously (IV) (into a vein in the arm).

Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. The study will last approximately 33 weeks excluding screening.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of 18.0 to 32.0 kilogram per square meter (kg/m²), inclusive

Part C and D Only:

* Have a body weight at least 50 kilograms and BMI within the range 18.0 to 40.0 kg/m² (inclusive) at screening
* Have a diagnosis of adult-onset RA for at least 3 months prior to screening

Exclusion Criteria:

Healthy Participants for SAD Part A and MAD Part B Only:

* Have a history or presence of cardiovascular, respiratory, hepatic, ophthalmological, renal, gastrointestinal, endocrine, hematological, neurological, or psychiatric disorders capable of significantly altering the absorption, metabolism, or elimination of drugs

Participants with RA for Parts C and D Only:

* Have Class 4 RA according to American College of Rheumatology (ACR) revised criteria
* Have a 12-lead electrocardiogram (ECG) abnormality at screening
* Have a current or recent acute active infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 33
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4213663 | Baseline up to Week 33
  PK: Cmax of LY4213663
PK: Area Under the Concentration Versus Time Curve (AUC) of LY4213663 | Baseline up to Week 33
  PK: AUC of LY4213663

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - GNP Research at Mark Jaffe, MD, Cooper City, Florida
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Oasis Clinical Research, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY4213663 in Healthy Participants and Participants With Rheumatoid Arthritis — https://trials.lilly.com/en-US/trial/668755